CLINICAL TRIAL: NCT04661683
Title: Investigating the Secondhand Effects of Hookah Smoking and Vaping
Brief Title: Secondhand Effects of Hookah (i.e., Waterpipe) Smoke and Aerosol
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Mary Rezk-Hanna, PhD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 20-001570
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-01

CONDITIONS: Hookah Smoking; Secondhand Aerosol; Vascular Stiffness; Vaping
MeSH Terms: conditions — Water Pipe Smoking; Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exposure to Combustible Hookah Smoke (Experimental): Participants will be exposed to combustible hookah smoke. To mitigate the impact of carryover effects, the exposure sessions will be separated by a minimum of 7-days.
  Interventions: Other: Combustible Hookah Smoke
- Exposure to Electronic Hookah Aerosol (Experimental): Participants will be exposed to electronic hookah aerosol. To mitigate the impact of carryover effects, the exposure sessions will be separated by a minimum of 7-days.
  Interventions: Other: Electronic Hookah Aerosol
- Exposure to Clean Air (Experimental): Participants will be exposed to Clean Room Air. To mitigate the impact of carryover effects, the exposure sessions will be separated by a minimum of 7-days.
  Interventions: Other: Clean Room Air

INTERVENTIONS:
Other: Combustible Hookah Smoke — Exposure to combustible hookah smoke for a duration of 60 minutes.
  Arms: Exposure to Combustible Hookah Smoke
Other: Electronic Hookah Aerosol — Exposure to electronic hookah aerosol for a duration of 60 minutes.
  Arms: Exposure to Electronic Hookah Aerosol
Other: Clean Room Air — Exposure to room air for a duration of 60 minutes.
  Arms: Exposure to Clean Air

SUMMARY:
In the United States, secondhand smoke is the third leading preventable cause of death. Flavored hookah (waterpipe) tobacco smoking, a highly social activity common in hookah bars, is a key source of SHS exposure. While smoke-free air laws have decreased exposure to secondhand smoke, the majority of laws do not include hookah smoking. Thus, as a social outlet for youth and young adults, hookah smoke exposure may harm non-smokers, including women of reproductive age or pregnant, hookah bar workers, children, and individuals with heart and lung disease. While more is known on the acute effects of active hookah smoking and the literature is emerging on active e-hookah vaping, little is known about the acute vascular effects of secondhand exposure to hookah smoke and aerosol. The study aims to examine the acute effects of secondhand exposure of hookah smoke and aerosol on endothelial and vascular function. Eligible volunteers will be invited to participate in a total of 3 study visits (2-3 hours each): e-hookah aerosol exposure, charcoal-heated hookah smoke exposure and smoke-free room air. Non-invasive blood pressure and blood flow measurements will be taken before and after the exposure sessions.

ELIGIBILITY:
Inclusion Criteria:

* 21-49 years old
* Never a smoker: do not use any tobacco products or nicotine delivery systems, including cigarettes, cigars (traditional and filtered), cigarillos, hookah, smokeless tobacco (i.e., loose snus, moist snuff, dip, spit, or chewing tobacco), pipe tobacco, snus pouches, dissolvable tobacco or vaping.
* no evidence of cardiopulmonary disease by history/physical
* blood pressure (BP) < 140/90 mmHg
* resting heart rate (HR) < 100 bpm
* BMI >18 or < 30kg•m2
* no prescription medication
* No exposure to environmental tobacco smoke for at least one week prior to the study date.

Exclusion Criteria:

* exhaled carbon monoxide >6 ppm
* (+) pregnancy test
* other conditions deemed unsafe to participate, such as breastfeeding

Ages: 21 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-06-25 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Flow-Mediated Dilation (FMD) | Pre- and post- the 60-minute exposure sessions
  Using ultrasound, FMD of the brachial artery induced by reactive hyperemia, will be used to measure endothelium-dependent vasodilator function. Baseline diameter and velocity will be recorded for 45 seconds and resumed 30 seconds before cuff deflation and continuously for 2 minutes after deflation to obtain true peak vasodilatory response.
Arterial stiffness | Pre- and post- the 60-minute exposure sessions
  Using applanation tonometry, pulse wave velocity will be used to measure cebtral arterial stiffness.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No